CLINICAL TRIAL: NCT03520881
Title: The Development and Pilot Testing of a Pediatric Algorithmic Software Tool to Help Manage Asthma (ASTHMA)-Educator
Brief Title: Pediatric ASTHMA-Educator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-2693A
Record Dates: First submitted 2018-04-13; First posted 2018-05-11 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: There is one group (intervention arm only) in this proof of concept study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric ASTHMA-Educator arm (Experimental): This arm corresponds to the pediatric version of the ASTHMA-Educator mobile application.
  Interventions: Other: Pediatric ASTHMA-Educator mobile application

INTERVENTIONS:
Other: Pediatric ASTHMA-Educator mobile application — This intervention represents a mobile application (accessible by iOS and Android devices) that provides asthma education through games and videos.

SUMMARY:
This project seeks to develop and pilot test the pediatric ASTHMA-Educator mobile application.

DETAILED DESCRIPTION:
This project seeks to develop and pilot test the pediatric ASTHMA-Educator mobile application. The study is being conducted at Montefiore Medical Center among pediatric (7-17 years old) patients with persistent asthma. We are collecting process and clinical outcomes in a longitudinal study design.

ELIGIBILITY:
Inclusion Criteria:

English-speaking individuals between 7-17 years with:

* Persistent asthma (diagnosis made by a healthcare provider) on a daily controller medication
* Able to give informed consent
* Smartphone (iOS or Android) access

Exclusion Criteria

* Use of oral corticosteroids in the 2 weeks prior to the baseline visit
* Pregnancy
* Severe psychiatric or cognitive problems that would prohibit an individual from understanding and completing the protocol
* Patients that previously received the ASTHMA-Educator application

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline asthma control to 2, 4, and 6 months | Baseline, 2 months, 4 months, 6 months
  Asthma symptom burden as measured by the Asthma Control Test

SECONDARY OUTCOMES:
Patient satisfaction measured by the Client Satisfaction Questionnaire-8 | Baseline, 2 months, 4 months, 6 months
  Patient satisfaction measured by the Client Satisfaction Questionnaire-8
Change from baseline asthma knowledge to 2 months, 4 months, 6 months | Baseline, 2 months, 4 months, 6 months
  Asthma knowledge as measured by the Asthma Knowledge Questionnaire
Asthma quality of life as measured by the Pediatric Asthma Impact Scale | Baseline, 2 months, 4 months, 6 months
  Patient's asthma quality of life measured by the Pediatric Asthma Impact Scale
Self-reported medication adherence | Baseline, 2 months, 4 months, 6 months
  Patients' self-reported medication adherence measured by the Medication Adherence Rating Scale
Asthma emergency department visits | Baseline, 2 months, 4 months, 6 months
  Asthma emergency department visits
Asthma hospitalizations | Baseline, 2 months, 4 months, 6 months
  Asthma hospitalizations
Asthma-related steroid courses | Baseline, 2 months, 4 months, 6 months
  Asthma-related steroid courses

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share aggregated and deidentified data in the form of abstracts and publications.
Supporting Information: SAP, CSR